CLINICAL TRIAL: NCT05444452
Title: Comparison Between Abluminal Biodegradable Polymer Ultrathin Sirolimus-eluting Stent and Durable-polymer Everolimus-eluting Stent (GENOSS Randomized Clinical Trial)
Brief Title: GENOSS Coronary Stent Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Genoss Company Limited, Suwon, Korea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENOSS
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Ischemic Heart Disease
Keywords: coronary stent; ischemic heart disease; acute coronary syndrome
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GENOSS stent arm (Experimental): Coronary lesions of the subjects this arm will be treated with GENOSS stent when in need of stent implantation
  Interventions: Device: Implanatation of Genoss DES sirolimus-eluting coronary system
- XIENCE stent arm (Active Comparator): Coronary lesions of the subjects this arm will be treated with Xience stent when in need of stent implantation
  Interventions: Device: Implanatation of Xience DES everolimus-eluting coronary system

INTERVENTIONS:
Device: Implanatation of Genoss DES sirolimus-eluting coronary system — Percutaneous coronary intervention will proceed as per clinical guidelines, under operator's discretion. Genoss stent will be implanted if the lesion is deemed necessary to be revascularized by stenting
  Arms: GENOSS stent arm
Device: Implanatation of Xience DES everolimus-eluting coronary system — Percutaneous coronary intervention will proceed as per clinical guidelines, under operator's discretion. Xience stent will be implanted if the lesion is deemed necessary to be revascularized by stenting
  Arms: XIENCE stent arm

SUMMARY:
This study aims to evaluate the efficacy and safety of abluminal biodegradable polymer ultrathin sirolimus-eluting stent (Genoss stent) as compared with a durable-polymer everolimus-eluting stent (Xience stent) in patients with coronary artery disease.

DETAILED DESCRIPTION:
After the introduction of the drug-eluting stents (DES), the rates of device-related failure or target lesion failure (TLF) such as restenosis has been markedly decreased, compared with the era of bare-metal stents. Nevertheless, the risk of ischemic events including very late stent thrombosis after percutaneous coronary intervention (PCI) has still remained even though the use of DES, presumably because of hypersensitivity to the polymer with persistent inflammation and delayed re-endothelialization. To overcome these issues, second-generation DES with thinner stent strut and biocompatible or biodegradable polymer were developed. Several trials demonstrated that second-generation DES provides more favorable outcome in comparison with first-generation DES. Especially, among second-generation DES, biodegradable polymer DES showed better ischemic outcomes compared to durable polymer DES in some studies.

Genoss DES™ (Genoss Company Limited, Suwon, Korea) is one of newer second-generation DESs with a cobalt-chromium platform with an abluminal biodegradable polymer containing sirolimus. The Genoss DES™ is the first Korean sirolimus-eluting stent on the market and it has ultrathin strut with 70 μm strut thickness with 3 μm thin abluminal polymer coating containing Sirolimus. The polymer is designed to release approximately 70% of the total drug amount within 30 days of the implantation and is entirely absorbable within 9 months. Thus, only the metal component of the stent will remain. In the first-in-man trial comparing Genoss DES™ and Promus Element™ stent (Boston Scientific Co., Natick, MA, USA), angiographic and clinical outcomes were similar at a 9-month follow-up. However, the study was too small to conclude that the Genoss DES™ is safe and efficient for de novo coronary stenosis. To date, there has been no large-scale randomized trial evaluating the safety and efficacy of Genoss DES™.

Therefore, the purpose of this trial is to determine the efficacy and safety of Genoss DES™ as compared with Xience everolimus-eluting stent (Abbott Vascular, Santa Clara, California, USA) which is widely used and has proven efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

① Subject must be at least 19 years of age

② Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.

③ Patients with stable coronary artery disease or acute coronary syndrome and at least one lesion with greater than 50% diameter stenosis suitable for stent implantation

Exclusion Criteria:

* Pregnant women ② Patients unable to provide consent, ③ Patients with known intolerance to aspirin, clopidogrel, ticagrelor, prasugrel, heparin or components of drug-eluting stents (sirolimus or everolimus)

  * Patients who have non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2022-04-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
TLF at 1 year | 1 year
  A composite of cardiac death, target vessel-MI, or clinically indicated TLR by percutaneous or surgical methods at 1 year

SECONDARY OUTCOMES:
TLF at 3 years | 3 years
  A composite of cardiac death, target vessel-MI, or clinically indicated TLR by percutaneous or surgical methods at 3 year
Target vessel failure | 1 and 3 years
  a composite of cardiac death, target vessel-MI, or clinically indicated target-vessel revascularization [TVR] by percutaneous or surgical methods at 1 and 3 years
All-cause death | 1 and 3 years
  All-cause death at 1 and 3 years
Cardiac death | 1 and 3 years
  Cardiac death at 1 and 3 years
MI | 1 and 3 years
  Myocardial infarction, as defined by the protocol of this study, at 1 and 3 years
Stent thrombosis | 1 and 3 years
  F. Stent thrombosis (definite or probable by Academic Research Consortium [ARC] definition) at 1 and 3 years
All-cause death or MI | 1 and 3 years
  All-cause death or MI at 1 and 3 years
Cardiac death or MI | 1 and 3 years
  Cardiac death or MI at 1 and 3 years
Cardiac death, MI or stent thrombosis | 1 and 3 years
  Cardiac death, MI or stent thrombosis at 1 and 3 years
Stroke | 1 and 3 years
  Stroke at 1 and 3 years
Clinically indicated TLR | 1 and 3 years
  Clinically indicated target lesion revascularization at 1 and 3 years
Clinically indicated TVR | 1 and 3 years
  Clinically indicated target vessel revascularization at 1 and 3 years
Any revascularization | 1 and 3 years
  Any revascularization at 1 and 3 years
Major bleeding | 1 and 3 years
  Major Bleeding (BARC [Bleeding Academic Research Consortium] types 3 or 5) at 1 and 3 years
Bleeding | 1 and 3 years
  Bleeding (BARC type 2, 3, or 5) at 1 and 3 years
Restricted mean survival time for the TLF | 1 and 3 years
  Restricted mean survival time for the TLF over 1 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Hyeon-Cheol, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No